CLINICAL TRIAL: NCT03267680
Title: A Two-Cohort, Open-label Phase 2 Trial of the IRX-2 Regimen in Women With Squamous Cervical Intraepithelial Neoplasia 3 (CIN 3) or Vulvar Intraepithelial Neoplasia 3 (VIN 3)
Brief Title: IRX-2 Regimen in Treating Women With Cervical Squamous Intraepithelial Neoplasia 3 or Squamous Vulvar Intraepithelial Neoplasia 3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Brooklyn ImmunoTherapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5GYN-16-2; NCI-2017-01402 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 5GYN-16-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Cervical Squamous Cell Carcinoma In Situ; Vulvar High Grade Squamous Intraepithelial Lesion
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Cyclophosphamide; Indomethacin; IRX 2; Geritol; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (IRX-2) (Experimental): Patients receive cyclophosphamide IV on day 1 and IRX-2 via submucosal injections in the cervix or SC for vulvar lesions on days 4-7. Patients also receive indomethacin PO TID, zinc-containing multivitamins PO QD and omeprazole PO on days 1-21. Treatment repeats every 6 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Beginning week 25, patients undergo surgical resection.
  Interventions: Drug: Cyclophosphamide; Drug: Indomethacin; Biological: IRX-2; Other: Laboratory Biomarker Analysis; Dietary Supplement: Multivitamin; Drug: Omeprazole; Procedure: Therapeutic Conventional Surgery
- Arm II (placebo) (Active Comparator): Patients receive cyclophosphamide IV on day 1 and placebo via submucosal injections in the cervix or SC for vulvar lesions on days 4-7. Patients also receive indomethacin PO TID, zinc-containing multivitamins PO QD and omeprazole PO on days 1-21. Treatment repeats every 6 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Beginning week 25, patients undergo surgical resection.
  Interventions: Drug: Cyclophosphamide; Drug: Indomethacin; Other: Laboratory Biomarker Analysis; Dietary Supplement: Multivitamin; Drug: Omeprazole; Other: Placebo; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
Drug: Indomethacin — Given PO
Biological: IRX-2 — Given via submucosal injection or SC
  Arms: Arm I (IRX-2)
Other: Laboratory Biomarker Analysis — Correlative studies
Dietary Supplement: Multivitamin — Given zinc-containing multivitamin PO
  Other Names: Geritol; Vitamin Supplements (NOS)
Drug: Omeprazole — Given PO
Other: Placebo — Given via submucosal injections or SC
  Other Names: placebo therapy; sham therapy
  Arms: Arm II (placebo)
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection

SUMMARY:
This randomized phase II trial studies how well an IRX-2 Regimen works in treating women with cervical squamous intraepithelial neoplasia 3 or squamous vulvar intraepithelial neoplasia 3. The IRX-2 Regimen consists of a single dose of cyclophosphamide, followed by 21 days of indomethacin, zinc-containing multivitamins, and omeprazole. IRX-2, a human cell-derived biologic with multiple active cytokine components, may act as an immune booster to stimulate the immune system. Giving cyclophosphamide and IRX-2 may work better at treating cervical squamous intraepithelial neoplasia or squamous vulvar intraepithelial neoplasia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the proportion of subjects who achieve a pathologic complete response (CR) or partial response (PR) in regimen 1 versus regimen 2 at week 25, based on the resected surgical specimen.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity and feasibility of administration of IRX-2 in subjects with confirmed cervical intraepithelial neoplasia (CIN) 3 or vulvar intraepithelial neoplasia (VIN) 3.

II. To evaluate multiple parameters to assess the activity of the IRX-2 regimen for the treatment of CIN 3 or VIN 3: the occurrence of clinical CRs or PRs at weeks 6, 13 and 25.

III. To evaluate multiple parameters to assess the activity of the IRX-2 regimen for the treatment of CIN 3 or VIN 3: frequency of elimination of human papillomavirus (HPV) in cervical or vulvar tissue using a commercial HPV genotyping assay and viral load determination by quantitative polymerase chain reaction (PCR).

IV. To evaluate multiple parameters to assess the activity of the IRX-2 regimen for the treatment of CIN 3 or VIN 3: analysis of the immune infiltrates in the resected surgical specimens.

V. To evaluate multiple parameters to assess the activity of the IRX-2 regimen for the treatment of CIN 3 or VIN 3: immunophenotypic analysis of peripheral blood lymphocytes.

VI. To evaluate multiple parameters to assess the activity of the IRX-2 regimen for the treatment of CIN 3 or VIN 3: frequency of serum antibodies to HPV E6, E7 and L1 proteins by enzyme-linked immunosorbent assay (ELISA).

VII. To evaluate multiple parameters to assess the activity of the IRX-2 regimen for the treatment of CIN 3 or VIN 3: ribonucleic acid (RNA) expression profiling of immune-inflammatory markers from post-treatment resected surgical specimens.

OUTLINE: Patients are randomized to 1 of 2 arms.

Arm I: Patients receive cyclophosphamide intravenously (IV) on day 1 and IRX-2 via submucosal injections in the cervix or subcutaneously (SC) for vulvar lesions on days 4-7. Patients also receive indomethacin orally (PO) three times daily (TID), zinc-containing multivitamins (PO) once daily (QD) and omeprazole orally (PO) on days 1-21.

Arm II: Patients receive cyclophosphamide IV on day 1 and placebo via submucosal injections in the cervix or SC for vulvar lesions on days 4-7. Patients also receive indomethacin PO TID, zinc-containing multivitamins PO QD and omeprazole PO on days 1-21.

In both arms, treatment repeats every 6 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Beginning week 25, patients undergo surgical resection.

After completion of study treatment, patients are followed up at 1-8 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous CIN 3, or VIN 3 (usual type only)
* The subject is either surgically sterile, postmenopausal, or agrees to practice an effective method of birth control as determined by the investigator (to be continued throughout the study period), except that subjects with CIN 3 are not permitted to use a cervical cap or diaphragm for contraception
* White blood cell > 2,500/ mcL (> 2.5 x 10^9/L)
* Absolute neutrophil count > 1,000/ microliter (> 1 x 10^9/L)
* Platelet count > 75,000/ mcL (> 75 x 10^9/L)
* Hemoglobin >= 8 g/dL (>= 80 g/L) (subjects who have received a transfusion or erythropoietin up to one week prior to receiving the first dose of cyclophosphamide are eligible for the study)
* International normalized ration (INR) or prothrombin time (PT) < 1.5 x ULN (upper limit of normal)
* Activated partial thromboplastin time (aPTT) < 1.5 x ULN
* Serum creatinine < 1.5 x ULN
* Total bilirubin < 2.0 x ULN unless thought to be related to inherited bilirubin conjugation disorder (ie Gilbert?s disease)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN
* The subject is geographically accessible for ongoing follow-up and is committed to comply with the designated visits
* The subject is capable of understanding and complying with the protocol and has signed the enrollment informed consent form at screening

Exclusion Criteria:

* For subjects with cervical dysplasia: evidence of atypical glandular cells or adenocarcinoma in situ (ACIS) based on cervical cytology, colposcopy or biopsy
* For subjects with either cervical or vulvar squamous dysplasia: evidence of microinvasive squamous carcinoma based on cytology, colposcopy or biopsy
* Pregnancy or lactation
* Allergy to ciprofloxacin or other quinolones (because ciprofloxacin is used in preparation of IRX-2)
* Allergy to indomethacin (a necessary component of the regimen) or to acetylsalicylic acid (aspirin) due to likely allergy cross-reaction
* Aldara (imiquimod) for the topical treatment of lower genital tract warts or dysplasia within 3 months of study enrollment
* Known to be positive for human immunodeficiency virus-1 (HIV-1) antibody, human immunodeficiency virus-2 (HIV-2) antibody, hepatitis B surface antigen, or hepatitis C virus antibody
* Known to have other immunodeficiency diseases, including cellular immunodeficiencies, hypogammaglobulinemia, or dysgammaglobulinemia
* Immunotherapy (eg, interferons, tumor necrosis factor, interleukins) or biological response modifiers (granulocyte-macrophage colony-stimulating factor, granulocyte colony-stimulating factor, macrophage colony-stimulating factor) or any investigational drug within 3 months of study enrollment
* Concurrent treatment with systemic corticosteroids at a dose of >= 5 mg/day of prednisone (or equivalent)
* Subjects should not take aspirin (except for low-dose aspirin as prescribed for vascular disease) or other non-prescribed, non-steroidal anti-inflammatory agents from randomization to surgery
* An infectious process or any other significant illness such as an autoimmune disease or advanced age that in the opinion of the investigator would compromise the subject?s ability to mount an immune response
* Impaired hepatic, renal or hematological function, evidenced by:

  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin >= 2 times upper limit of normal (ULN),
  * Serum creatinine >= 2 times ULN, or
* Clinically significant active cardiovascular disease, including a history of myocardial infarction within the past 6 months, heart failure as defined by New York Heart Association classes III or IV, and/or blood pressure greater than 160/90 mm Hg (1 repeat measure allowed no more than 5 minutes after the first measurement)
* History of severe allergic reaction to insect bites or stings, or to any biologic pharmaceutical product, including compounds similar to the test article
* Any medical contraindications, allergies or previous therapy that would preclude treatment with the components of the IRX-2 regimen, i.e., cyclophosphamide, indomethacin, zinc-containing multivitamins or omeprazole
* Donation or loss of > 450 mL of blood or plasma within 30 days of randomization

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2024-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Roman, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Oklahoma Health Sciences Center, Stephenson Cancer Center, Oklahoma City, Oklahoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began recruiting in November 2017 and recruitment ended in August 2023. All participants were seen and treated at USC Norris Comprehensive Cancer Center and/or at LAC+USC Medical Center.
Period: Overall Study
Arm/Group | Arm I (IRX-2) | Arm II (Placebo)
Started (Arm I patients CIN3 = 6 VIN3 = 1) | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (IRX-2) | Arm II (Placebo) | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 3 | 10
Smoking Status [Count of Participants; unit: Participants]
  Never Smoke | 4 | 1 | 5
  Former Smoker | 3 | 1 | 4
  Current Smoker | 0 | 1 | 1
Alcohol Use [Count of Participants; unit: Participants]
  Yes | 4 | 1 | 5
  No | 3 | 2 | 5
HPV Status (High Risk Positive) [Count of Participants; unit: Participants] | 7 | 3 | 10
Ever Received HPV Vaccine [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 5 | 2 | 7
  Unknown | 1 | 1 | 2
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 5 | 2 | 7
  Postmenopausal | 2 | 0 | 2
  Surgical/Other for Amenorrhea | 0 | 1 | 1
Number of Pregancies [Count of Participants; unit: Participants]
  0 | 2 | 1 | 3
  1 or 2 | 3 | 1 | 4
  2 or more | 2 | 1 | 3
Number of Abortions/Miscarriages [Count of Participants; unit: Participants]
  0 | 4 | 3 | 7
  1 | 3 | 0 | 3
Number of Still Births [Count of Participants; unit: Participants]
  0 | 7 | 2 | 9
  Unknown | 0 | 1 | 1
Number of Live Births [Count of Participants; unit: Participants]
  0 | 3 | 1 | 4
  1 or 2 | 2 | 1 | 3
  2 or more | 2 | 0 | 2
  Unknown | 0 | 1 | 1
Currently Sexually Active [Count of Participants; unit: Participants]
  No | 2 | 1 | 3
  Yes | 4 | 2 | 6
  Unknown | 1 | 0 | 1
Number of Lifetime Partners [Count of Participants; unit: Participants]
  1 or 2 | 2 | 0 | 2
  2 or more | 1 | 2 | 3
  Unknown | 4 | 1 | 5
Contraception Use [Count of Participants; unit: Participants]
  No | 2 | 1 | 3
  Yes | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response
Description: Complete Response (CR) is defined as absence of intraepithelial neoplasia, Partial Response (PR) is defined as a lower grade of dysplasia than present at baseline (for example, grade 3 decreasing to grade 1).
Time Frame: Week 25
Population: All patients who received at least 1 cycle is included. There is no statistical analysis performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (IRX-2) | Arm II (Placebo)
Number analyzed (Participants) | 7 | 3
Participants
  Pathologic Complete Response | 1 | 1
  Persistent CIN3/VIN3 | 6 | 2

2. Secondary Outcome: Incidence of Adverse Events of IRX-2 Administration
Description: Will be assessed by the incidence and severity of adverse events, serious adverse events, as classified and graded according to the current version of the Common Terminology Criteria for Adverse Events version 4.
Time Frame: Up to 30 months
Population: All treated patients are included
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (IRX-2) | Arm II (Placebo)
Number analyzed (Participants) | 7 | 3
Participants
  Grades 1 and 2 Adverse Events | 7 | 3
  Grades 3 and 4 Adverse Events | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Arm I (IRX-2) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (IRX-2) (N=7) | Arm II (Placebo) (N=3)
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Mucositis Oral (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 6 | 2
Injection Site Reaction (General disorders) | 2 | 1
Pain (General disorders) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 0
White Blood Cell Decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal Inflammation (Reproductive system and breast disorders) | 1 | 0
Vaginal Pain (Reproductive system and breast disorders) | 2 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 2
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Burning in Clitoris (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT03267680/Prot_SAP_000.pdf